CLINICAL TRIAL: NCT01874171
Title: Determination of Epidermal Growth Factor Receptor-inhibitor (Cetuximab) Versus Standard Chemotherapy (Cisplatin) Early And Late Toxicity Events in Human Papillomavirus-positive Oropharyngeal Squamous Cell Carcinoma
Brief Title: Determination of Cetuximab Versus Cisplatin Early and Late Toxicity Events in HPV+ OPSCC
Acronym: De-ESCALaTE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Warwick (Other)
Collaborators: Cancer Research UK (Other); University of Birmingham (Other); University of Oxford (Other)
Responsible Party: Principal Investigator, Prof. Janet Dunn, Professor of Clinical Trials, University of Warwick
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMRCT0034; 2011-005165-21 (EudraCT Number); ISRCTN33522080 (Other: ISRCTN)
Record Dates: First submitted 2013-06-06; First posted 2013-06-10 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Oropharyngeal Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cisplatin (Active Comparator): Three doses of cisplatin 100mg/m2 given at days 1, 22 and 43 from start of radiotherapy.
  Interventions: Drug: Cisplatin
- Cetuximab (Experimental): Initial dose of 400mg/m2 one week before start of radiotherapy followed by seven weekly doses of 250 mg/m2 during radiotherapy.
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Cisplatin
  Arms: Cisplatin
Drug: Cetuximab
  Arms: Cetuximab

SUMMARY:
Oropharyngeal squamous cell carcinoma (OPSCC) incidence is increasing rapidly in the developed world. This has been attributed to a rise in Human Papillomavirus (HPV) infection. HPV+OPSCC is considered a distinct disease entity, affecting younger patients and has a good prognosis following treatment. Subsequently, patients can live with the considerable side effects for several decades.

Radiotherapy and cetuximab (Epidermal Growth Factor Receptor-inhibitor) have demonstrated similar efficacy to 'platin' chemoradiotherapy (current standard treatment containing platinum-based compounds) in head and neck cancer, but is potentially less toxic.

Results of this trial will be used to determine the optimum treatment of this debilitating cancer, with the primary aim of decreasing toxicity and improving quality of life for HPV+OPSCC patients.

ELIGIBILITY:
Inclusion Criteria:

* American Joint Committee on Cancer (AJCC) TNM Stage III-IVa (T3N0-T4N0, and T1N1-T4N3) oropharyngeal squamous cell carcinoma (SCC) tumours
* Clinical multidisciplinary team decision to treat with primary curative cisplatin chemoradiotherapy
* No previous treatment including surgery, except node biopsies or diagnostic tonsillectomy
* Medically fit (ECOG 0, 1 or 2)
* Adequate cardiovascular, haematological, renal and hepatic function
* Age > 18 years
* Written informed consent given
* Using adequate contraception [male and female participants]. Must take contraceptive measures during, and for at least six months after treatment.

Exclusion Criteria:

* Distant metastasis (i.e. AJCC TNM stage IVc disease)
* AJCC TNM Stage T1-2N0 disease
* Treated with primary radical surgery to the primary site (e.g. resection)
* Concurrent use of CYP3A4 inducers or inhibitors. [A standard course of dexamethasone or aprepitant for the prevention of cisplatin-induced nausea and vomiting is permitted]
* Serious cardiac illness or other medical conditions precluding the use of cisplatin or cetuximab [no history of clinically significant cardiac disease, serious arrhythmias, or significant conduction abnormalities; no uncontrolled seizure disorder; no active neurologic disease; no neuropathy greater than grade 1]
* Patients who have p16+ tumours who also have N2b, N2c or N3 nodal disease and whose lifetime smoking history is also more than 10 pack years (i.e. have both risk factors).
* Pregnant or lactating
* Previous treatment for any other cancer with cytotoxics, radiotherapy or anti-EGFR therapies
* Inadequate renal, haematological or liver functions [Absolute neutrophil count <1,500/mm3; platelet count <100,000/mm3; WBC <3,000/mm3; haemoglobin <9 g/dL. [Haemoglobin correction by transfusion permitted.] Bilirubin > 1.5 times upper limit of normal (ULN); alkaline phosphatase > 2.5 times ULN; AST and ALT > 2.5 times ULN. Creatinine > 1.5 mg/dL; Creatinine clearance < 60 mL/min]
* Patients with clinically significant hearing impairment
* Life expectancy less than 3 months
* Other malignancy within the past 3 years except basal cell skin cancer or pre-invasive carcinoma of the cervix.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2012-11-15 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Compare severe (acute and late) toxicity (Grade 3-5) caused by cetuximab and radiotherapy to that caused by cisplatin and radiotherapy. | Up to two years after end of treatment.

SECONDARY OUTCOMES:
Overall number of events of acute severe toxicity between treatment arms. | Up to and including three months after end of treatment.
Overall number of events of late severe toxicity between treatment arms. | From three months up to two years after end of treatment.
Quality of life outcomes assessed by EORTC QLQ C30 and HN35 between the two treatment arms. | Baseline, end of treatment, and 3, 6, 12 & 24 months after end of treatment.
Effect on swallowing of the two treatment arms (assessed by MDADI and by PEG or RIG utilisation rate at 1 and 2 years). | Baseline, end of treatment, and 3, 6, 12 & 24 months after end of treatment.
Cost-effectiveness of the two treatment arms (assessed by EuroQoL-5D). | Up to two years after end of treatment.
  Questionnaires completed at the following time points: Baseline, end of treatment, and 3, 6, 12 & 24 months after end of treatment.
Overall survival and recurrence between the two arms. | Up to two years after end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hisham Mehanna, PhD, BMedSc (hons), FRCS, Study Chair — University of Birmingham
Locations (33):
- Ireland (2):
  - St Luke's Hospital, Dublin
  - Beaumont Hospital, Dublin
- VU University Medical Center, Amsterdam, Netherlands
- United Kingdom (30):
  - Aberdeen Royal Infirmary, Aberdeen
  - Royal United Hospital, Bath
  - Clatterbridge Cancer Centre, Bebington
  - Bradford Royal Infirmary, Bradford
  - Bristol Haematology & Oncology Centre, Bristol
  - Velindre Hospital, Cardiff
  - Cheltenham General Hospital, Cheltenham
  - Colchester General Hospital, Colchester
  - Castle Hill Hospital, Cottingham
  - University Hospitals Coventry & Warwickshire, Coventry
  - Royal Derby Hospital, Derby
  - Queen Elizabeth Hospital Birmingham, Edgbaston
  - Western General Hospital, Edinburgh
  - Royal Devon & Exeter Hospital, Exeter
  - Royal Surrey County Hospital, Guildford
  - St James's Institute of Oncology, Leeds
  - Leicester Royal Infirmary, Leicester
  - University College Hospital, London
  - Royal Marsden Hospital, London
  - James Cook University Hospital, Middlesbrough
  - New Cross Hospital, New Cross
  - Northampton General Hospital, Northampton
  - Norfolk & Norwich University Hospital, Norwich
  - Nottingham University Hopsital, Nottingham
  - Glan Clwyd Hospital, Rhyl
  - Weston Park Hospital, Sheffield
  - Royal Shrewsbury Hospital, Shrewsbury
  - Royal Marsden Hospital, Sutton
  - Singleton Hospital, Swansea
  - Musgrove Park Hospital, Taunton

REFERENCES:
- See also: De-ESCALaTE study website — http://www.warwick.ac.uk/go/deescalate